CLINICAL TRIAL: NCT02743078
Title: Phase II Trial Of Optune® Plus Bevacizumab In Bevacizumab-Refractory Recurrent Glioblastoma
Brief Title: Optune® Plus Bevacizumab in Bevacizumab-Refractory Recurrent Glioblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Treatment now available commercially
Sponsor: RTOG Foundation, Inc. (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 3503; RF 3503 (Other: RTOG Foundation)
Record Dates: First submitted 2016-04-05; First posted 2016-04-19 (Estimated); Results first posted 2020-11-17 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2020-10

CONDITIONS: Glioblastoma; Glioma; Gliosarcoma
Keywords: Glioblastoma; Glioma; Gliosarcoma; Optune; TTFields
MeSH Terms: conditions — Glioblastoma; Glioma; Gliosarcoma | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Bevacizumab and TTFields Therapy (Experimental): Bevacizumab starts on the first day (+/- 1 day) of Tumor Treating Fields (TTFields) therapy. Treatment is given until disease progression or the development of adverse events that require complete discontinuation.
  Interventions: Drug: Bevacizumab; Device: TTFields Therapy

INTERVENTIONS:
Drug: Bevacizumab — 10 mg/kg every 2 weeks intravenously over 30 minutes.
  Other Names: Avastin
Device: TTFields Therapy — Device is worn continuously at least 18 hours a day on average, with 1-3 days off every four weeks.
  Other Names: Optune; Tumor Treating Fields Therapy; TTF Therapy

SUMMARY:
This phase II trial will investigate the efficacy and safety of the addition of Optune (Tumor Treating Fields [TTFields] Therapy) to bevacizumab for patients with bevacizumab-refractory recurrent glioblastoma.

DETAILED DESCRIPTION:
Patients that have recurrent glioblastoma that has progressed on bevacizumab continue to receive bevacizumab with the addition of Tumor Treating Fields Therapy. Treatment is given until disease progression or the development of adverse events that require complete discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of glioblastoma or other grade IV malignant glioma (including variants of glioblastoma i.e., gliosarcoma, giant cell glioblastoma, etc.).
* Confirmation of tumor recurrence or progression on contrast magnetic resonance imaging (MRI) (with and without gadolinium contrast) as determined by Response assessment in neuro-oncology (RANO) criteria within 14 days prior to registration for patients who did not have recent resection of their glioblastoma or only had a stereotactic biopsy.
* Patients having undergone recent resection (within 5 weeks prior to registration) of their glioblastoma to treat current recurrence prior to study treatment must have recovered from the effects of surgery (including patient's skin having fully recovered from the surgical wound) Note: a 4-week window is required after surgery prior to starting treatment. For central nervous system (CNS) -related stereotactic biopsies, a minimum of 7 days must have elapsed prior to registration.
* Residual disease of recurrent glioblastoma is not mandated for eligibility into the study. To best assess the extent of residual disease post-operatively, a post-operative MRI scan must be performed prior to registration and is recommended to be within 96 hours post-surgery (although 24-48 hours would be optimum). Note: Patients who did have surgery with a post-operative contrast-enhanced scan falling outside the 5-week window prior to registration, must have a repeat MRI scan within 14 days prior to registration.
* Patients with up to two recurrences are allowed.
* Failure on bevacizumab (either as a monotherapy or a combination) as most recent regimen confirmed by tumor recurrence on MRI.

  * The patient must have failed no more than one regimen of bevacizumab.
  * The patient must not have received bevacizumab as an upfront treatment in newly diagnosed glioblastoma.
  * There must be a minimum of 14 days (i.e., an interval equal to or greater than 14 days) since last treatment with bevacizumab and registration
* History/physical examination within 14 days prior to registration
* Karnofsky performance status ≥ 70 within 14 days prior to registration
* Age ≥ 22
* Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3
* Platelets ≥ 75,000 cells/mm3
* Hemoglobin (Hgb) ≥ 9.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 9.0 g/dl is acceptable.)
* Creatinine ≤ 1.5 mg/dl
* Urine protein: creatinine (UPC) ratio < 1.0 within 14 days prior to registration OR urine dipstick for proteinuria ≤ 2+ (patients discovered to have > 2+ proteinuria on dipstick urinalysis at baseline must have a UPC ratio done that is <1.0 to be eligible. If the UPC ratio is ≥ 1.0 then the patients should undergo a 24-hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).

  *Note: UPC ratio of spot urine is an estimation of the 24-hour urine protein excretion; a UPC ratio of 1 is roughly equivalent to a 24-hour urine protein of 1 gm. UPC ratio is calculated using one of the following formulas:
  * [urine protein]/[urine creatinine]: if both protein and creatinine are reported in mg/dL
  * [(urine protein) x0.088]/[urine creatinine]: if urine creatinine is reported in mmol/L
* Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN) within 14 days prior to registration
* Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 3.0 x ULN within 14 days prior to registration
* Patients on full dose anticoagulants (e.g., warfarin or low molecular weight (LMW) heparin) must meet both of the following criteria:

  1. No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices) within 14 days prior to registration
  2. One of the below criteria must be met based on patient's therapy:

     1. Warfarin: In-range international normalized ratio (INR) (usually between 2 and 3) within 14 days prior to registration
     2. LMW heparin or novel oral anti-coagulant: stable dose within 14 days prior to registration
* Patients must have recovered from the toxic effects of prior therapy at the time of registration as follows:

  * 28 days from the administration of any investigational agent
  * 28 days from administration of prior cytotoxic therapy with the following exceptions:

    * 14 days from administration of vincristine or irinotecan
    * 42 days from administration of nitrosoureas
    * 21 days from administration of procarbazine
  * 7 days from administration of non-cytotoxic agents [e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count)]

    * Female patients of child-bearing potential must have a negative serum pregnancy test within 14 days prior to registration.
    * Patient must be maintained on a stable or decreasing dose of corticosteroid for at least 5 days before the baseline scan.
    * Minimum interval since completion of radiation treatment at the time of registration is 90 days.
    * Patient must provide study specific informed consent prior to study entry.

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years. (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible).
* Infra-tentorial tumor.
* > 1 cm diameter of blood seen on contrast MRI (with and without gadolinium contrast)
* Major surgery such as intra-thoracic, intra-abdominal or intra-pelvic (with the exception of craniotomy), open biopsy or significant traumatic injury ≤ 4 weeks prior to registration, or patients who have had minor procedures, percutaneous biopsies or placement of vascular access device ≤ 1 week prior to registration, or who have not recovered from side effects of such procedure or injury.
* Implanted pacemaker, defibrillator or deep brain stimulator, other implanted electronic devices in the brain.
* Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months prior to registration.
* Transmural myocardial infarction within the last 6 months prior to registration
* Cerebrovascular accident (CVA), transient ischemic attack (TIA) within the last 6 months prior to registration
* Pulmonary embolism (PE) within the last 6 months prior to registration
* Uncontrolled hypertension (defined by a systolic blood pressure (SBP) ≥ 160 mm Hg or diastolic blood pressure (DBP) ≥ 100 mm Hg while on anti-hypertensive medications) within 14 days prior to registration.
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration.
* Chronic lung disease or Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration.
* Severe hepatic disease, defined as a diagnosis of Child-Pugh Class B or C hepatic disease.
* Known HIV positive patients.
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g. active or uncontrolled infection, uncontrolled diabetes) that could cause unacceptable safety risks or compromise compliance with the protocol.
* Skull defects such as missing bone flap, a shunt, or bullet fragments.
* Significant intracranial pressure as per treating physician that may require surgical intervention.
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception.
* Breast feeding women.
* Prior allergic reaction to bevacizumab or severe adverse event with bevacizumab.
* Known sensitivity to conductive hydrogels.
* Prior treatment with the Optune® system.
* Active treatment on another clinical trial.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manmeet Ahluwalia, MD, FACP, Principal Investigator — RTOG Foundation
Locations (11):
- United States (11):
  - University of California, San Diego, La Jolla, California
  - University of California Irvine, Chao Family Comprehensive Cancer Center, Orange, California
  - Miami Cancer Institute at Baptist Health, Miami, Florida
  - UF Health Cancer Center at Orlando Health, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Washington University School of Medicine, St Louis, Missouri
  - University of Rochester, Rochester, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab and TTFields Therapy
Started | 3
Eligible Populaton | 3
Eligible With Six-month Follow-up Data | 3
Completed (Participants contributing data to results are considered to have completed the study) | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab and TTFields Therapy
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 55 [34 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at 6 Months
Description: Number of participants alive at 6 months. Out of the planned 80 eligible patients, if 36 or more were alive at six months then the null hypothesis that the six-month survival rate is 35% or less would be rejected, concluding that the six-month survival is at least 35%. No testing was done due to the small number of participants resulting from early study closure.
Time Frame: From registration to six months
Population: Eligible with six-month follow-up data
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab and TTFields Therapy
Number analyzed (Participants) | 3
Participants | 1

2. Secondary Outcome: Overall Survival (OS)
Description: Survival time is defined as time from registration the to date of death from any cause or last known follow-up (censored) and was to be estimated by the Kaplan-Meier method. Given the small number of participants due to early study closure, only the number of patients last reported to be alive at time of study termination is reported.
Time Frame: From registration to study termination. Maximum follow-up was 21.8 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab and TTFields Therapy
Number analyzed (Participants) | 3
Participants | 1

3. Secondary Outcome: Progression-Free Survival
Description: Progression is defined by the Modified Response Assessment in Neuro-Oncology (RANO) Response Criteria. (The precise definition is too long to be included here.) Progression-free survival time is defined as time from registration to the date of first progression, death, or last known follow-up. Progression-free survival rates were to be estimated using the Kaplan-Meier method. Given the small number of participants due to early study closure, only the number of patients last reported to be alive without progression at time of study termination is reported.
Time Frame: From registration to study termination. Maximum follow-up was 21.8 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab and TTFields Therapy
Number analyzed (Participants) | 3
Participants | 0

4. Secondary Outcome: Number of Participants With Partial or Complete Response
Description: Modified Response Assessment in Neuro-Oncology (RANO) Response Criteria was used to define response and progression. (The precise definitions are too long to be included here.) Objective response is defined as complete or partial response. The percentage of participants with objective response was to be estimated using the exact binomial method with accompanying 95% confidence intervals. Given the small number of participants due to early study closure, only the number of patients with objective response is reported.
Time Frame: From registration to study termination. Maximum follow-up was 21.8 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab and TTFields Therapy
Number analyzed (Participants) | 3
Participants | 0

5. Secondary Outcome: Number of Participants With Grade 3+ Treatment-related Adverse Events
Description: Adverse events were graded using the Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Grade refers to the severity of the adverse event (AE). The CTCAE v4.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to AE. The percentage of participants with grade 3 or higher treatment-related adverse events was to be estimated using the exact binomial method with accompanying 95% confidence intervals.
Time Frame: From registration to study termination. Maximum follow-up was 21.8 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab and TTFields Therapy
Number analyzed (Participants) | 3
Participants | 2

ADVERSE EVENTS:
Time Frame: Every 28th day during treatment, at progression, then every 8 weeks for one year, then every 12 weeks for one year, then every 6 months. Maximum follow-up at time of study termination was 21.8 months.
Arm/Group | Bevacizumab and TTFields Therapy
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab and TTFields Therapy (N=3)
Intracranial hemorrhage (Nervous system disorders) | 1
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab and TTFields Therapy (N=3)
Fatigue (General disorders) | 1
Pain (General disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Dysphasia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3

LIMITATIONS AND CAVEATS:
This study stopped accrual early due to unmet targeted accrual goals with 3 subjects accrued out of 85 planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT02743078/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT02743078/ICF_001.pdf